CLINICAL TRIAL: NCT02075749
Title: Comparison of Triamcinolone Acetonide Mucoadhesive Film With Liquorice Mucoadhesive Film On Radiotherapy-Induced Oral Mucositis: A Randomized Double-Blinded Clinical Trial
Brief Title: Comparing Triamcinolone Acetonide Mucoadhesive Films With Licorice Mucoadhesive Films
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mehdi Nasr Isfahani, Dr. Nasr, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 393009
Record Dates: First submitted 2014-02-26; First posted 2014-03-03 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Mucositis
Keywords: irradiation; mucositis; triamcinolone acetonide; licorice; mucoadhesive film
MeSH Terms: conditions — Mucositis | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- triamcinolone acetonide mucoadhesive (Active Comparator): 30 patients received triamcinolone acetonide mucoadhesive films
  Interventions: Drug: Triamcinolone Acetonide
- Licorice (Experimental): 30 patients received licorice mucoadhesive films
  Interventions: Drug: licorice mucoadhesive films
- Mucoadhesive film (Placebo Comparator): 30 patients received mucoadhesive films without any drug ingredients

INTERVENTIONS:
Drug: Triamcinolone Acetonide
  Other Names: made in Germany (Merck)
  Arms: triamcinolone acetonide mucoadhesive
Drug: licorice mucoadhesive films — 30 patients received licorice mucoadhesive films
  Other Names: AFTOGEL Patch
  Arms: Licorice

SUMMARY:
Abstract:

Background: Complementary and alternative medicine (CAM) had proven efficacy in pain relief, correction of nutritional status and improving the performance status. However, lack of standardization is the major obstacle for any scientific evaluation of any CAM trial. Mucositis is a major complication of irradiation in head and neck (H&N) tumors, the addition of chemotherapy to irradiation may enhance this dose limiting problem. Licorice is a strong demulcent that had been effectively used in treatment of peptic ulcer. The main purpose of this study was to compare the therapeutic safety and efficacy of T. and L. mucoadhesive films on oral mucositis in terms of pain control and/or ulcer treatment.

Methods and Materials: the study was a double-blind, randomized prospective trial of two types of mucoadhesive films in the management of oral mucositis occurred during head and neck cancer ( HNC ) radiotherapy. oral mucositis was assessed using a quantitative scale (WHO scales) and symptoms were assessed using visual analogue scales (VAS). 60 patients were enrolled in the study; there were 30 patients in the Triamcinolone (T) and 30 in the Licorice (L) group. In the T- group, patients received triamcinolone acetonide mucoadhesive films containing 1mg of the drug and patients in the L- group received licorice mucoadhesive films, an herbal agent. Data were collected at baseline, then twice a week for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* men and nonpregnant women
* women of childbearing age who were non-pregnant by pregnancy test and and using medically prescribed contraceptive
* no previous radiation therapy applied in the head and neck
* medically fit for a course of radical radiotherapy
* an ability to remain in the study for its entire duration

Exclusion Criteria:

* pregnant women
* women of childbearing potential in whom medically prescribed birth control was not used
* concurrent chemotherapy
* history of heavy alcohol or drug abuse judged to be important by the investigator - concomitant therapy with an investigational drug, or cancer chemo therapeutics or immunosuppressive medications
* sensitivity or intolerance to triamcinolone or licorice, lactose or similar formulations
* inability to provide informed consent
* actively bleeding gastric ulcer, severe esophageal reflux
* major surgery, trauma or burns in the preceding 4 weeks
* clinically significant hepatic, neurologic, endocrine, or other systemic disease-making implementation of the protocol or results difficult.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-05; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
pain score | 4 weeks
  at the end of each consecutive week the pain score was recorded.

SECONDARY OUTCOMES:
mucositis grade | 4 weeks
  the grading of mucositis was assessed and recorded at the end of each week.

OTHER OUTCOMES:
quality of life | 4 weeks
  patient's satisfaction and ability to perform social activity were assessed at the end of trial.

CONTACTS AND LOCATIONS:
Locations (1):
- Omid ( or Sayyed-O-Shohada) Hospital, Isfahan, Isfahan, Iran